CLINICAL TRIAL: NCT01333553
Title: Monitoring the Response of Port Wine Stain Birthmarks to Laser Therapy With Wide-field
Brief Title: Monitoring the Response of Port Wine Stain Birthmarks to Laser Therapy With Wide-field Functional Imaging Technologies
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Bernard Choi, Ph.D., Assistant Professor Biomedical Engineering, University of California, Irvine
Other Study IDs: 20107376
Record Dates: First submitted 2010-08-03; First posted 2011-04-12 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: PORT WINE STAIN
Keywords: birthmark
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Image-guided remove Port Wine Stain: Image-guided surgery remove Port Wine Stain
  Interventions: Device: Image-guided remove Port Wine Stain

INTERVENTIONS:
Device: Image-guided remove Port Wine Stain — Image-guided surgery remove Port Wine Stain

SUMMARY:
The researcher develop non-invasive imaging modalities for assessment of port wine stain during laser therapy treatment of Port Wine Stain. The imaging modalities will be used to guide immediate retreatment of regions of persistent perfusion during the procedure.

DETAILED DESCRIPTION:
The researcher can use imaging system operates by projecting low-power near-infrared structured light patterns on to the tissue of interest in a non-contact, reflection geometry and then capturing the reflectance with a camera.The system can image the depth-resolved optical properties of in-vivo tissues, allowing rapid, non-invasive visualization of sub-surface structures of Port Wine Stain.

ELIGIBILITY:
Inclusion Criteria:

* All minors, birth to 18 years of age or older with Port Wine Stain birthmark
* Ability to understand and carry out subject instructions
* Sign photograph release form

Exclusion Criteria:

* Inability to understand and/or carry out instructions
* Pregnant women
* Do not sign photograph release form

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be selected from an outpatient population with Port Wine Stain birthmark at Beckman Laser Institute and Medical Clinic, University of California, Irvine. Patients with Port Wine Stain birthmark will be candidates for participation.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2010-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Image-guided surgery remove Port Wine Stain | 24 hours
  Image-guided surgery remove Port Wine Stain

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Choi, PhD, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute Medical clinic, Irvine, California, United States